CLINICAL TRIAL: NCT01161225
Title: Peer-Assisted Asthma Self-Management Program for Adolescents
Brief Title: Teen Asthma Project
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Hyekyun Rhee, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R21NR009837 (NIH)
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Asthma
Keywords: Adolescents; Peer leader program; asthma camp; asthma control; quality of life; self-efficacy; knowledge; attitudes; barrier perceptions
MeSH Terms: conditions — Asthma; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peer-led asthma self-managment program (Experimental)
  Interventions: Behavioral: Peer-assisted asthma self-management program
- Adult-led asthma self-management program (Active Comparator)
  Interventions: Behavioral: Adult-led asthma self-management program

INTERVENTIONS:
Behavioral: Peer-assisted asthma self-management program — Intervention group: An asthma self-management program (Power Breathing™) was implemented by trained peer leaders at an asthma day camp. The program consisted of 3 sessions (appx. 45-60 min/session): basic asthma education (pathophysiology, triggers); psychosocial issues of asthma; and asthma self-management (peak flow monitoring and medication). The program was delivered by trained peer leaders paired for each small group of 6-8 teens. Group activities involved discussion, strategic thinking, knowledge-testing games and role plays.
  Arms: peer-led asthma self-managment program
Behavioral: Adult-led asthma self-management program — Control group: The group attended an adult-led day camp where 2 NPs and a MD offered didactic asthma education based on the Power Breathing™ program.
  Arms: Adult-led asthma self-management program

SUMMARY:
Aims of this study are:

1. To determine the feasibility of implementing the intervention using a peer-assisted asthma day camp for adolescents with asthma.
2. To determine patterns of change in knowledge, attitudes toward asthma, self-efficacy, perception of barriers, and self-management behaviors, asthma control and quality of life over time among peer leaders.
3. To test the following hypothesis:

   * Adolescents participating in a peer-assisted asthma camp program will report improved knowledge, attitudes toward asthma, self-efficacy, and self-management behaviors, decreased perception of barriers, and increased asthma control and quality of life at 3-, 6- and 9-months post-intervention compared with the adult-led camp group.
4. To examine the moderating effect of personal factors (e.g., age, sex, socioeconomic status, race, illness status, family support) on intervention outcomes such as self-management behaviors, asthma control and quality of life in adolescents with asthma.
5. To examine the effect of the peer-assisted camp program on self-reported health care utilization including emergency department visits, days of hospitalization, outpatient visits by comparing between baseline and 9-months post-camp data and between the peer-led camp and the adult-camp programs.

ELIGIBILITY:
Inclusion Criteria:

1. age between 13-18 years
2. mild, moderate or severe persistent asthma specified by the NHLBI Asthma guidelines
3. asthma diagnosis > 1 year
4. no other major chronic/emotional health concerns
5. ability to understand spoken and written English. Participants were recruited from the communities through flyers, newspaper ads, and referrals from clinics and schools.

Eligibility criteria for peer leaders included:

1. age between 16-20 years
2. nomination from school teachers/nurses or health care providers
3. average grade point B or above in the past school year
4. fulfillment of eligibility criteria (2)-(5) prescribed for adolescent participants.

Exclusion Criteria:

* learning disabilities based on reports from parents, teachers or clinicians

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyekyun Rhee, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Background] Rhee H, Ciurzynski SM, Yoos HL. Pearls and pitfalls of community-based group interventions for adolescents: lessons learned from an adolescent asthma cAMP study. Issues Compr Pediatr Nurs. 2008 Jul-Sep;31(3):122-35. doi: 10.1080/01460860802272888. PMID 18728958
- [Result] Rhee H, Belyea MJ, Ciurzynski S, Brasch J. Barriers to asthma self-management in adolescents: Relationships to psychosocial factors. Pediatr Pulmonol. 2009 Feb;44(2):183-91. doi: 10.1002/ppul.20972. PMID 19142893
- [Result] Rhee H, Belyea MJ, Elward KS. Patterns of asthma control perception in adolescents: associations with psychosocial functioning. J Asthma. 2008 Sep;45(7):600-6. doi: 10.1080/02770900802126974. PMID 18773334
- [Result] Rhee H, McQuillan BE, Belyea MJ. Evaluation of a peer-led asthma self-management program and benefits of the program for adolescent peer leaders. Respir Care. 2012 Dec;57(12):2082-9. doi: 10.4187/respcare.01488. PMID 22710616
- [Result] Rhee H, Pesis-Katz I, Xing J. Cost benefits of a peer-led asthma self-management program for adolescents. J Asthma. 2012 Aug;49(6):606-13. doi: 10.3109/02770903.2012.694540. Epub 2012 Jul 4. PMID 22758599
- [Result] Rhee H, Belyea MJ, Hunt JF, Brasch J. Effects of a peer-led asthma self-management program for adolescents. Arch Pediatr Adolesc Med. 2011 Jun;165(6):513-9. doi: 10.1001/archpediatrics.2011.79. PMID 21646583
- [Result] Rhee H, Belyea MJ, Halterman JS. Adolescents' perception of asthma symptoms and health care utilization. J Pediatr Health Care. 2011 Mar-Apr;25(2):105-13. doi: 10.1016/j.pedhc.2009.10.003. PMID 21320682

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: This is the group who participated in a peer-led asthma self-management program. This group attended an asthma self-management program led by peer leaders in a camp setting. Afterward, the group received monthly phone contacts from their peer leaders who offered continuous support, encouragement and reminder throughout the 9-month study period. Follow-up assessments (including quality of life, asthma control, healthcare utilization, asthma knowledge, self-efficacy and attitude toward asthma) were completed every 3 months for 9 months.
- Control Group: This is the group who participated in an adult-led asthma self-management program. This group attended an asthma self-management program offered by healthcare professionals (physician and nurse practitioner) in a camp setting. Follow-up assessments (including quality of life, asthma control, healthcare utilization, asthma knowledge, self-efficacy and attitude toward asthma) were completed every 3 months for 9 months.
- Peer Leader Group: Teens who participated in the study as peer leaders. This group attended 3-day intense training program (a total of 12 hours) offered by a nurse practitioner. The training program covered not only asthma-related content but also leadership training. Then, each peer leader pair facilitated the peer-led asthma self-management program for a small group of 6-8 teens in the camp and made monthly contacts for 9 months. Follow-up assessments (including quality of life, asthma control, healthcare utilization, asthma knowledge, self-efficacy and attitude toward asthma) were completed every 3 months for 9 months.
Period: Overall Study
Arm/Group | Intervention Group | Control Group | Peer Leader Group
Started | 59 | 53 | 14
Completed | 45 | 44 | 12
Not Completed | 14 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Peer Leader Group | Total
Number analyzed (Participants) | 59 | 53 | 14 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.31 (1.36) | 14.97 (1.29) | 18.28 (1.90) | 15.50 (1.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 11 | 75
  Male | 26 | 22 | 3 | 51
Region of Enrollment [Number; unit: participants]
  United States | 59 | 53 | 14 | 126

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Asthma Quality of Life Questionnaire (PAQLQ)
Description: Twenty-three items cover problems identified as being most important and troublesome in children's everyday lives due to asthma. This scale is effective in evaluating and discriminating because of its high sensitivity to changes in asthma status within and between individuals with varying severity of asthma. Respondents are asked to recall impairments experienced during the previous week. The scale consists of three subdomains including symptoms (10 items), emotional function (8 items) and activity limitation (5 items). Each item was measured on a 7-point scale; 1 indicates maximum impairment, and 7 indicates no impairment. Higher total scores indicate better levels of functioning. Total scores were computed by summing responses from all items (range:24-161)
Time Frame: 9 months post camp
Population: The number of participants analyzed includes only those who stayed in the study and completed the 9-months assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group | Peer Leader Group
Number analyzed (Participants) | 43 | 41 | 9
units on a scale | 140.30 (21.04) | 125.12 (25.95) | 138.11 (16.44)

2. Primary Outcome: Asthma Control Questions
Description: This measure assesses the frequencies of the limitation of daily activity, asthma symptoms (daytime and nighttime) and use of rescue medication in the past 4 weeks on a 5-point scale (0-4). Total summed scores were computed (range: 4-16). Higher total scores indicate better controlled asthma.
Time Frame: 9 months post camp
Population: the number of participants analyzed includes only those who stayed in the study and completed the 9-months assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group | Peer Leader Group
Number analyzed (Participants) | 43 | 41 | 9
units on a scale | 14.84 (1.86) | 14.19 (1.83) | 14.89 (1.05)

3. Secondary Outcome: Asthma Self-Efficacy
Description: This 14-item scale was developed to measure the child's confidence in attack prevention (e.g., learn asthma self-management skills, correct use of medication) and attack management (e.g., control symptoms, decide which medication to use). Total summed scores were computed (range: 21-70). Higher total scores indicate greater degree of self-efficacy.
Time Frame: 9 months post camp
Population: the number of participants analyzed includes only those who stayed in the study and completed the 9-months assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group | Peer Leader Group
Number analyzed (Participants) | 43 | 41 | 9
units on a scale | 56.19 (10.02) | 51.93 (9.09) | 57.44 (3.84)

4. Secondary Outcome: Illness Management Survey
Description: This 29-item scale was developed to assess perception of barriers and to predict risk for poor self-management in adolescents with chronic illness. This scale categorizes barriers based on internal processes (e.g., cognitive skills, denial, pessimistic thinking) and contextual forces (e.g., illness-related factors, peer/family influences). Total summed scores were computed (range: 28-91). Higher scores indicate the high levels of perceived barriers to self-management.
Time Frame: 9 months post camp
Population: the number of participants analyzed includes only those who stayed in the study and completed the 9-months assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group | Peer Leader Group
Number analyzed (Participants) | 43 | 41 | 9
units on a scale | 56.74 (16.95) | 64.61 (13.11) | 60.55 (10.31)

5. Secondary Outcome: Attitude Toward Illness Scale
Description: This 13-item scale was designed to assess children's attitude toward their health condition. The scale includes questions such as "how good or bad do you feel it is that you have ___?" and, "how often do you feel that your ___ is your fault?" Respondents answer each question on a 5-point Likert-type scale (1-5). Total summed scores (range: 25-65) was constructed to reflect respondents' overall attitudes. Higher scores indicated positive attitudes.
Time Frame: 9 months post camp
Population: the number of participants analyzed includes only those who stayed in the study and completed the 9-months assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group | Peer Leader Group
Number analyzed (Participants) | 43 | 41 | 9
units on a scale | 50.05 (7.30) | 47.12 (794) | 45.44 (5.90)

6. Secondary Outcome: Asthma Knowledge Questionnaire
Description: This 30-item instrument was developed to measure children's knowledge on triggers and symptom identifications, and asthma management procedures (i.e., what to do and how to do it) in a true/false format. Total scores (range: 14-30) were computed by summing the number of items correctly answered. The higher scores indicate greater knowledge levels.
Time Frame: 9 months post camp
Population: the number of participants analyzed includes only those who stayed in the study and completed the 9-months assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group | Peer Leader Group
Number analyzed (Participants) | 43 | 41 | 9
units on a scale | 25.86 (3.11) | 25.02 (3.57) | 28.11 (1.45)

7. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) % Predicted
Description: Maximal amount of air one can forcefully exhale in one second. It is then converted to a percentage of normal. Range: 55-124 for the current sample.
Time Frame: 9 months post camp
Population: the number of participants analyzed includes only those who stayed in the study and completed spirometry at 9-months assessment.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Groups:
- Intervention Group: This is the group who participated in a peer-led asthma self-management program.
- Control Group: This is the group who participated in an adult-led asthma self-management program
- Peer Leader Group: Teens who participated in the study as peer leaders
Arm/Group | Intervention Group | Control Group | Peer Leader Group
Number analyzed (Participants) | 36 | 39 | 9
percentage of predicted FEV1 | 100.77 (13.75) | 97.67 (11.03) | 102.11 (16.04)

8. Secondary Outcome: Health Care Utilization Events
Description: Participants report the following information for the prior 3-month period; their emergency department visits for asthma; hospitalization for asthma; urgent office visit for worsening asthma; routine office visit; specialist visit. A cumulative number of events were computed by adding # of visits and # of days (for hospitalization) occurred in the past 3 months .
Time Frame: 9-months postcamp
Population: the number of participants analyzed includes only those who stayed in the study and completed the 9-months assessment.
Measure: Mean (Standard Deviation); unit: average number of events
Arm/Group | Intervention Group | Control Group | Peer Leader Group
Number analyzed (Participants) | 43 | 41 | 9
average number of events | 0.53 (1.12) | 0.78 (1.27) | 0.77 (1.28)

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group | Peer Leader Group
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/53 | 0/14
Other Adverse Events (participants affected / at risk) | 0/59 | 0/53 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No